CLINICAL TRIAL: NCT04425941
Title: Artificial Intelligence Based Colorectal Polyp Histology Prediction by Using Narrow-band Imaging Magnifying Colonoscopy
Brief Title: Polyp Artificial Intelligence Study
Status: Completed | Type: Observational
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PetzACTHospital
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Software Analysis on Polyp Histology Prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: artificial intelligence diagnosis — artificial intelligence prediction of colorectal polyp histology

SUMMARY:
Background We are developing artificial intelligence based polyp histology prediction (AIPHP) method to automatically classify Narrow Band Imaging (NBI) magnifying colonoscopy images to predict the non-neoplastic or neoplastic histology of polyps.

Aim Our aim was to analyse the accuracy of AIPHP and NICE classification based histology predictions and also to compare the results of the two methods.

Methods We examined colorectal polyps obtained from colonoscopy patients who had polypectomy or endoscopic mucosectomy. Polyps detected by white light colonoscopy were observed then by using NBI at the optical maximum magnificent (60x). The obtained and stored NBI magnifying images were analysed by NICE classification and by AIPHP method parallelly. Pathology examinations were performed blinded to the NICE and AIPHP diagnosis, as well. Our AIPHP software is based on a machine learning method. This program measures five geometrical and colour features on the endoscopic image.

ELIGIBILITY:
Inclusion Criteria:

* endoscopic diagnosis of colorectal polyp

Exclusion Criteria:

* colonoscopy result without polyps or IBD diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptoms of colorectal polypoid laesions, colorectal cancer screening patients
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Software accuracy of polyp histology prediction | 2014-2020
  Artificial intelligence software diagnosis in comparison with the polyp histology